CLINICAL TRIAL: NCT01838967
Title: A Randomized, Open-label, Single Dosing, Three-way Crossover Clinical Trial to Investigate the Pharmacokinetic Drug-drug Interaction of Cilnidipine 10 mg and Valsartan 160 mg After Oral Administration in Healthy Male Volunteers
Brief Title: A Drug Interaction Study of Cilnidipine and Valsartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID_IDCV_1301
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: cilnidipin and valsartn; pharmacokinetic drug drug interaction; oral administration; healthy male subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- C - V - C+V (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: C - V - C+V
- V - C - C+V (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: V - C - C+V
- V - C+V - C (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: V - C+V - C
- C+V - V - C (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: C+V - C - V
- C+V - C - V (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: C+V - V - C
- C - C+V - V (Experimental): C - Cilnidipine 10mg will be administered orally only one time. V - Valsartan 160mg will be administered orally only one time. C+V - Cilnidipine 10mg plus Valsartan 160mg will be administered orally only one time
  Interventions: Drug: C - C+V - V

INTERVENTIONS:
Drug: C - V - C+V — Drug will be administered to according to C - V - C+V sequence for 3 period.
  Arms: C - V - C+V
Drug: C - C+V - V — Drug will be administered to according to C - C+V - V sequence for 3 period.
  Arms: C - C+V - V
Drug: V - C - C+V — Drug will be administered to according to V - C - C+V sequence for 3 period.
  Arms: V - C - C+V
Drug: V - C+V - C — Drug will be administered to according to V - C+V - C sequence for 3 period.
  Arms: V - C+V - C
Drug: C+V - C - V — Drug will be administered to according to C+V - C - V sequence for 3 period.
  Arms: C+V - V - C
Drug: C+V - V - C — Drug will be administered to according to C+V - V - C sequence for 3 period.
  Arms: C+V - C - V

SUMMARY:
The investigators investigate the potential pharmacokinetic drug-drug interaction between Cilnidipine 10 mg and Valsartan 160 mg in healthy male volunteers who receive Cilnidipine 10 mg alone, Valsartan 160 mg , and both together in a 3 period repeatedly.

DETAILED DESCRIPTION:
To evaluate the safety, drug-tolerance, pharmacokinetics of Cilnidipine 10 mg or Valsartan 160 mg monotherapy or Cilnidipine 10 mg and Valsartan 160 mg combination in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 20 to 40 years
2. The result of Body Mass Index(BMI) is not less than 18.5 kg/m2 , no more than 25 kg/m2 and body weight are least 55 kg
3. Subjects who have no congenital or chronic disease and no abnormal symptom or opinion
4. Acceptable serum test, hematologic test, blood chemistry examination, urin test and ECG, physical examination during screening
5. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. A subject with clinical evidence or history of hepatic (including carrier of hepatitis virus), renal, respiratory, endocrine, neurologic, immunologic, hematologic, oncologic, psychiatric, or cardiovascular disease
2. A subject with a history of gastrointestinal disease or surgery (except simple appendectomy or repair of hernia), which can influence the absorption of the study drug
3. A subject with history of drug allergies (aspirin, antibiotics, including study drug etc.), or history of clinically significant allergies
4. Systolic blood pressure <100mmHg or Diastolic blood pressure < 60 mmHg, systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100mmHg(Sitting blood pressure) during the screening procedure.
5. Presence or history of drug abuse or positive result in urine drug screening test
6. Use any prescriptive medication, Korean traditional medication not considered acceptable by the clinical investigator during the last 14 days period before first dosing, or use any OTC medication not considered acceptable by the clinical investigator during the last 7 days period before first dosing (if used medication is considered acceptable by investigator, patients can be included)
7. Participation in clinical trials of any drug within 60 days prior to the participation of the study
8. Blood donation during 2 months or apheresis during 1 month before the study
9. Use of alcohol over 21 units/weeks
10. Smoker who smoke more than 20 cigarettes per day
11. A subject who takes grapefruit, grapefruit juice, or grapefruit-containing products within 3 days prior to the participation of the study
12. A subject who takes St John's wort or some food including the ingredient within 14 days prior to the participation of the study
13. Judged to be inappropriate for the study by the investigator after reviewing clinical laboratory results or other reasons.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-04; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cmax of Cilnidipine 10 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
Cmax of Valsartan 160 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
AUClast of Cilnidipine 10 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
AUClast of Valsartan 160 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose

SECONDARY OUTCOMES:
Tmax of Cilnidipine 10 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
Tmax of Valsartan 160 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
AUCinf of Cilnidipine 10 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
CL/F of Cilnidipine 10 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
AUCinf of Valsartan 160 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose
CL/F of Valsartan 160 mg | 1d(8d, 15d) pre-dose, 0.5, 1, 2, 2.5, 3, 4, 5, 6, 8, 12, 24h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Sang You, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Jongno-gu, Seoul, South Korea